CLINICAL TRIAL: NCT06852079
Title: Safety & Efficacy of Qurs e Fishar in Mild to Moderate Hypertensive Patients in Pakistan
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Abdul Bari (Other)
Collaborators: Hamdard University (Other)
Responsible Party: Sponsor-Investigator, Abdul Bari, Co-Principal Investigator, Hamdard University
Organization: Hamdard University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-HLWP
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: HTN; Hypertension; Qurs e Fishar
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Effect of Qurs e Fishar on Hypertension (Experimental)
  Interventions: Other: Qurs e Fishar

INTERVENTIONS:
Other: Qurs e Fishar — Qurs e Fishar is a herbal remedy for Hypertension

SUMMARY:
The herbal medicine Qurs-e-Fishar to treat mild to moderate High blood pressure or hypertension comprises of Rauwolfia serpentina. A product of Hamdard Laboratories (Waqf) Pakistan.

A Phase III Safety & Efficacy Open-label, Single-Arm, Interventional, Multicenter, Study in mild to moderate hypertensive, adults (30 to 60 years of age) prescribed with study product for 12 weeks (84 days).

Primary End Points:

1. Reduction in diastolic blood pressure less than 130 / 80 mmHg at the end of the study period (accepted by WHO) or if there was a fall of 20 / 10 mmHg or more in diastolic blood pressure as compared to baseline.
2. Type, frequency and severity of ADRs during the study period.

Secondary End Points:

1. Compliance of the prescribed study medication.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign ICD
* Participant(s) are willing and able to fulfill the requirements of the study protocol
* Mild to moderate hypertensive
* Mild hypertension range (140-159/90-99 mm Hg)
* Moderate hypertension range (160-179/100-109 mm Hg)
* Be between the age of 30 to 60 year

Exclusion Criteria:

* Patients with recent history of following will be excluded:

  * Severe hypertension,
  * Congestive cardiac failure,
  * Left ventricular failure,
  * Myocardial ischemia,
  * Renal failure or
  * Cerebrovascular accidents

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 12 weeks
  Blood pressure (in mmHg) will be measure at baseline and again at first follow-up (4th week), than at second follow-up (at 8th week) the end of treatment (12th week).

CONTACTS AND LOCATIONS:
Locations (1):
- Taj Medical Complex, Hamdard University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No